CLINICAL TRIAL: NCT04561427
Title: Cohort Study on Sleep Architecture and Regulation, Cognitive Performance and Metabolism in Children With Narcolepsy
Brief Title: Pediatric Cohort Study
Acronym: COSACM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: COSACM_2020
Record Dates: First submitted 2020-08-27; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-08

CONDITIONS: Narcolepsy in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Patients with narcolepsy: * Patients between 0 and 18 years old
  * Patients diagnosed with primary or secondary narcolepsy
  * From both gender
  Interventions: Other: Study of Sleep architecture in children with narcolepsy

INTERVENTIONS:
Other: Study of Sleep architecture in children with narcolepsy — Evaluate the cognitive performances, the effects of narcolepsy treatments on sleep architecture and the metabolic status of these children

SUMMARY:
Narcolepsy is a rare disease that affects 0.05% of the general population. It is characterized by a dysregulation of the sleep wake regulation that leads to uncontrolled sleep episode during day and a disorganized sleep during night. These symptoms are due to a loss of hypocretin neurons in the brain leading to an inability to maintain wake properly. The physiopathology of this rare disease still needs investigations. Since we are a reference center for this disease, we propose to use patients files to better describe and document the sleep characteristics of these children, the cognitive performances, the effects of narcolepsy treatments on sleep architecture and the metabolic status of these children.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 0 and 18 years old
* Patients diagnosed with primary or secondary narcolepsy
* From both gender

Exclusion Criteria:

* Patients diagnosed with another sleep disorder
* Healthy patients
* Patients older than 18 years old

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children or adolescents (0 to 18 years old)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Sleep period (SP) evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In minutes
Total sleep time (TST) evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In minutes
Stage 1 duration evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In minutes
Stage 2 duration evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In minutes
Stage 3 duration evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In minutes
Stage 1 percentage evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In minutes
Stage 2 percentage evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In minutes
Stage 3 percentage evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In minutes
REM duration evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In minutes
REM percentage of TST evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In percentage of TST
Sleep efficiency evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  TST / SP in percentage
Sleep latency evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In minutes, first epoch of NREM or REM sleep
REM latency evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In minutes, first epoch of REM sleep from sleep onset
Wake after sleep onset (WASO) duration evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In minutes between sleep onset and sleep offset,
Micro-arousal index evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  Number of event / hour
Arousal index evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
Leg movements index evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  Number of event / hour
Apnea-hypopnea index evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  Number of respiratory events / hour
Mean saturation during sleep evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In percentage
Minimal saturation during sleep evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In percentage
Duration of SaO2<90% evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In percentage of total sleep time
Index of desaturation > 3% evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  Number of event / hour
Maximal CO2 during non-REM sleep evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In mmHg
Maximal CO2 during REM sleep evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In mmHg
Sleep time with PCO2 > 50 mmHg / TST evaluated by polysomnography (PSG) | During the 72 hours of the diagnostic' hospitalization
  In percentage
Sleep latency evaluated during multiple sleep latency test (MSLT) | During the 72 hours of the diagnostic' hospitalization
  In minutes
Stage 1 latency evaluated during multiple sleep latency test (MSLT) | During the 72 hours of the diagnostic' hospitalization
  In minutes
REM latency evaluated during multiple sleep latency test (MSLT) | During the 72 hours of the diagnostic' hospitalization
  In minutes
SOREM evaluated during multiple sleep latency test (MSLT) | During the 72 hours of the diagnostic' hospitalization
  In minutes
Power in frequency bands delta, alpha, gamma, theta evaluated during PSG | During the 72 hours of the diagnostic' hospitalization
Mean Bedtime evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  during week-end days and week days
Mean Wake up time evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  during week-end days and week days
Mean Time in bed evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  during week-end days and week days
Mean Total Sleep time evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  during week-end days and week days
Mean Waking time evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  during week-end days and week days
Mean Sleep period evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  during week-end days and week days
Mean Sleep efficiency evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  In percentage, during week-end days and week days
Mean wake after sleep onset duration evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  during week-end days and week days
Mean Sleep latency evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  during week-end days and week days
Mean fragmentation index evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  In percentage, during week-end days and week days
Mean Immobile time evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  In minutes, during week-end days and week days
Mean Moving time evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  In minutes, during week-end days and week days
Mean Number of immobile phases evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  during week-end days and week days
Mean Number of one minute immobility periods evaluated by actimetry | During 15 days before the diagnostic' hospitalization
  during week-end days and week days
Intellectual Quotient evaluated by the WISC | During the 72 hours of the diagnostic' hospitalization
  by a neuropsychologist.
Attention evaluated by the BLAST | During the 72 hours of the diagnostic' hospitalization
  during neuropsychological evaluation
Insomnia severity evaluated by Insomnia Severity Index (ISI) | During the 72 hours of the diagnostic' hospitalization
Depressive feelings evaluated by the Children Depression Inventory (CDI) | During the 72 hours of the diagnostic' hospitalization
Attention disorders symptoms evaluated by the Conners rating scale | During the 72 hours of the diagnostic' hospitalization
Fatigue evaluated by the Fatigue scale | During the 72 hours of the diagnostic' hospitalization
Estimated severity of the disease evaluated by the Severity scale | During the 72 hours of the diagnostic' hospitalization
Sleepiness evaluated by the Epworth sleepiness scale for children | During the 72 hours of the diagnostic' hospitalization
Sleepiness evaluated by the Karolinska scale | During the 72 hours of the diagnostic' hospitalization
Histamine rate in the cerebro-spinal fluid (CSF) , evaluated by lumbar punction | During the 72 hours of the diagnostic' hospitalization
  In pg/mL
Circadian typology evaluated by the Horne and Ostberg questionnaire | During the 72 hours of the diagnostic' hospitalization
Body fat evaluated by DEXA | During the 72 hours of the diagnostic' hospitalization
  In percentage
Lean mass evaluated by DEXA | During the 72 hours of the diagnostic' hospitalization
  In percentage
Leptin evaluated by blood test | During the 72 hours of the diagnostic' hospitalization
  In ng/ml
Total ghrelin evaluated by blood test | During the 72 hours of the diagnostic' hospitalization
Acylated ghrelin evaluated by blood test | During the 72 hours of the diagnostic' hospitalization
  In pg/mL
Non-acylated ghrelin ghrelin evaluated by blood test | During the 72 hours of the diagnostic' hospitalization
  In pg/mL
Fastin blood sugar evaluated by blood test | During the 72 hours of the diagnostic' hospitalization
  In mmol/L
Fasting insulin evaluated by blood test | During the 72 hours of the diagnostic' hospitalization
  In mUI/L,
Hba1C evaluated by blood test | During the 72 hours of the diagnostic' hospitalization
  In percentage
TSH evaluated by blood test | During the 72 hours of the diagnostic' hospitalization
  In mUI/L
T3 evaluated by blood test | During the 72 hours of the diagnostic' hospitalization
  In pmol/L
T4 evaluated by blood test | During the 72 hours of the diagnostic' hospitalization
  In pmol/L
Total cholesterol by blood test | During the 72 hours of the diagnostic' hospitalization
  In mmol/L
LDL by blood test | During the 72 hours of the diagnostic' hospitalization
  In mmol/L
HDL by blood test | During the 72 hours of the diagnostic' hospitalization
  In mmol/L
Triglycerides by blood test | During the 72 hours of the diagnostic' hospitalization
  In mmol/L
NFS by blood test | During the 72 hours of the diagnostic' hospitalization
Ionogram by blood test | During the 72 hours of the diagnostic' hospitalization
Epstein Barr Virus antibodies by serology | During the 72 hours of the diagnostic' hospitalization
  Positivity
Hepatitis B antibodies by serology | During the 72 hours of the diagnostic' hospitalization
  Positivity
Streptococcus antibodies by serology | During the 72 hours of the diagnostic' hospitalization
  Positivity
HLA evaluated by genotyping | During the 72 hours of the diagnostic' hospitalization
  Presence of the known HLA factor of predisposition for narcolepsy,
Urinary prolactin evaluated by urine test | During the 72 hours of the diagnostic' hospitalization
Urinary sulfatoxy-melatonin evaluated by urine test | During the 72 hours of the diagnostic' hospitalization
Urinary cortisol evaluated by urine test | During the 72 hours of the diagnostic' hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- : Sleep pediatric unit , Woman Mother Child Hospital, Hospices Civils de Lyon, Lyon, France